CLINICAL TRIAL: NCT06916429
Title: The Effectiveness of Psychological Interventions for Common Mental Disorders (EPIC): A Randomized Waitlist-controlled Superiority Trial.
Brief Title: The Effectiveness of Psychological Interventions for Common Mental Disorders
Acronym: EPIC
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Copenhagen (Other)
Collaborators: the Danish Psychological Association (Unknown); The Danish Regions: Foundation for Medical Research (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: IP-EC-19012024-1
Record Dates: First submitted 2025-03-31; First posted 2025-04-08 (Actual); Last update posted 2025-10-06 (Actual); Status verified 2025-04

CONDITIONS: Common Mental Disorders and/or Stress Related Symptoms
Keywords: psychotherapy; common mental disorders; depression; anxiety; randomized controlled trial
MeSH Terms: conditions — Depression; Anxiety Disorders | interventions — Psychotherapy; Psychosocial Intervention; Waiting Lists; Therapeutics

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Wailist Control Group (Other): Description: Clients in the waitlist control group will be placed on a waiting list for psychotherapy with treatment starting approximately four and a half months after the date of randomization.
  Objective: To serve as a control group to the intervention group receiving psychotherapy and to investigate distinct symptom trajectories during the waiting period.
  Interventions: Other: Waiting List for Psychotherapeutic Treatment
- Psychotherapy Intervention Group (Experimental): Description: Clients in the psychotherapy intervention group will receive psychotherapeutic treatment with treatment starting within 14 days of the randomization date.
  Objective: To determine the effectiveness of psychotherapy in the Danish primary sector over approximately a four-month period.
  Interventions: Other: Psychotherapeutic treatment

INTERVENTIONS:
Other: Psychotherapeutic treatment — The psychotherapeutic treatment will reflect the therapy practices that characterize the Danish primary sector.
  Treatment: Clients are referred by their GP to receive up to 12 individual psychotherapy sessions, typically of 50-60 minutes' duration. For clients with depression and anxiety as referral reason, it is possible to get a supplementary referral by the GP ensuring 12 more sessions, totaling 24 sessions of therapy.
  Procedure: Due to the Danish primary sector having relative freedom in method of choice, the psychologist carries out the psychotherapy according to the treatment principles they consider the most relevant, without clauses regarding specific models of therapy or manualization. The therapists register the therapeutic approaches and interventions used in each course of therapy on The Multitheoretical List of Therapeutic Interventions (MULTI-30)at the end of each treatment.
  Other Names: psychological treatment; psychotherapy; psychological intervention
  Arms: Psychotherapy Intervention Group
Other: Waiting List for Psychotherapeutic Treatment — Treatment: During the waiting list period, clients will not receive any psychotherapeutic treatment for their mental health issues in the Danish primary sector. However, their general practitioner may refer them to appropriate psychiatric treatment if their mental condition worsens and requires immediate treatment.
  Procedure: Clients in the waiting list group will fill in questionnaires on their symptom development during the waiting period. They will complete the same set of predictor and outcome questionnaires as the psychotherapy group.
  Other Names: waitlist; waiting list control group; waitlist for therapy
  Arms: Wailist Control Group

SUMMARY:
The primary aim of "the Effectiveness of Psychological Interventions for Common mental disorders" (EPIC) randomized controlled trial is to investigate whether a significantly larger symptom improvement is observed after approximately four months of psychotherapeutic treatment in the Danish primary sector compared to in a waiting list control group. The secondary aim of the study is to identify specific client and therapy characteristics that may predict the effectiveness of the therapy or the symptom development in the waiting list control group. The main hypothesis of the EPIC trial is:

1) Four and a half months after randomization, we will find a significantly lower level of symptoms on the primary outcome measure (PHQ-ADS) among clients who receive psychotherapy, compared to clients in the waiting list control group. In addition, we hypothesize to find significantly better outcomes in the psychotherapy group on all secondary outcome measures, four and a half months after randomization.

Researchers will compare:

* Psychotherapy starting within 14 days after the randomization date with
* Placement on a waiting list for psychotherapy with treatment starting approximately four and a half months after the randomization date

to investigate whether a larger symptom improvement is observed in the group receiving psychotherapy compared to the waiting list control group.

Participants will:

* Be referred by their general practitioner (GP) for publicly subsidized psychotherapy treatment in the primary care sector in Denmark, based on one of 11 referral reasons.
* Complete the baseline questionnaire containing background information, the primary and secondary outcome measures, and predictor questionnaires, and subsequently be randomized to either psychotherapy beginning within two weeks or a waiting list control group.
* Receive a brief symptom questionnaire (the PHQ-ADS) every other week after the randomization date via an SMS-based solution provided by REDCap.
* Complete the primary and secondary outcome measures approximately four and a half, eight and a half, and 16 and a half months after the randomization date.

DETAILED DESCRIPTION:
Aims:

The primary aim of this randomized controlled trial is to investigate whether a significantly higher symptom improvement is observed after approximately four months of psychotherapeutic treatment in the Danish primary sector compared to a waiting list control group. A supplementary aim is to explore whether the treatment effect is maintained during follow-up assessed approximately eight and 16 months after the beginning of treatment. The secondary aim of the study is to investigate whether specific client and therapy characteristics predicting the effect of the therapy and the symptom change in the waitlist control group can be identified, and whether the quality of the therapeutic alliance measured after approximately five weeks of therapy is related to the outcome of therapy.

The hypotheses of the study are as follows:

1. Four and a half months after randomization, we will find a significantly lower level of symptoms on the primary outcome measure (PHQ-ADS) among clients who receive psychotherapy, compared to clients in the waiting list control group. In addition, we hypothesize to find significantly better outcomes in the psychotherapy group on all secondary outcome measures, four and a half months after randomization.
2. We expect that the client's coping strategies, emotion regulation strategies, and level of personality pathology will be significantly related to symptom change and treatment dropout amongst the clients receiving psychotherapy, and to symptom change in the waitlist group, four and a half months after randomization.
3. We expect that the quality of the working alliance after approximately five weeks of therapy will be significantly related to symptom change on the PHQ-ADS after four and a half months of therapy. Conversely, we do not expect that the therapeutic orientation of the psychologist will be independently related to symptom change after four and a half months of therapy.
4. We will explore whether the symptom change observed after approximately four and a half months persists eight and a half and 16 and a half months after the beginning of therapy.

   Primary Analysis:

   - The primary analysis of the general treatment effect in the practice sector will consist of a multilevel longitudinal regression model. This model will assess the difference in the rate of change between the intervention group and the control group in the PHQ-ADS scores over a period of approximately four months of therapy.

   Secondary Analyses:
   * As a secondary analysis of the treatment effect, a multilevel logistic regression model will compare the difference in reliable remission rates on the PHQ-9 and the GAD-7 between the intervention group and the control group after approximately four months of therapy. The reliable remission rates on the PHQ-9 and the GAD-7 are employed by the IAPT in the UK and the PMHC in Norway, enabling us to benchmark our results with other studies examining the impact of psychotherapy in primary sectors similar to Denmark.
   * Another secondary analysis of the treatment effect will compare differences between the intervention group and the control group after approximately four months of therapy on the secondary continuous outcome measures, specifically the SPS, the CPS, the WHO-5, and the NEQ (see Measures).
   * Finally, in a secondary analysis of the treatment effect at follow-up, multilevel regression models will compare the pre-post change in the treatment group approximately eight and 16 months after the beginning of therapy with the change found after four months, and multilevel logistic regression models will compare the reliable remission rates on the PHQ-9 and the GAD-7 found at eight and 16 months with the rate found after approximately four months.

   Secondary Predictor Analyses:
   * In addition, we will conduct multilevel longitudinal regression models using the predictor variables (i.e., the client's sociodemographic and clinical characteristics, coping strategies, emotion regulation strategies, and level of personality pathology) as fixed effect predictors. The dependent variable will be the rate of change in the PHQ-ADS, measured in both arms of the trial after approximately four months of therapy. Moreover, we will conduct multilevel logistic regression analyses and repeat the predictor analyses in both arms of the study, using the treatment dropout rate as a binary dependent variable.
   * Moreover, a multilevel regression model on the association between the client-rated working alliance after approximately five weeks of therapy and the rate of change in the PHQ-ADS after approximately four months of therapy is conducted. In this analysis, the change score on the PHQ-ADS from treatment start to the fifth therapy week will be included as a covariate.

   All analyses are conducted as intention-to-treat with multiple imputations of missing data.

   Study Design:

   The study is designed as a pragmatic randomized controlled trial with a block randomization of clients referred by their general practitioner (GP) for psychotherapy treatment in the primary care sector in Denmark. The clients are randomized in a 1:1 allocation ratio to one of the following options:
   * Psychotherapy starting within 14 days of the randomization date
   * Placement on a waiting list for psychotherapy, with treatment starting four and a half months after the randomization date.

   Participants:

   Participants will typically be referred by their GP based on one of 11 referral reasons, which include:
   * Victims of traffic and other accidents
   * Relatives of seriously mentally ill persons
   * Persons suffering from a seriously debilitating illness
   * Relatives of persons suffering from a seriously debilitating illness
   * Relatives of recently deceased persons
   * Persons who have attempted suicide
   * Women having undergone an induced abortion after the 12th week of pregnancy
   * Persons who, before the age of 18, have been victims of incest or other sexual assaults
   * Persons aged 18 or above with mild to moderate depression
   * Persons aged 18 or above with mild to moderate anxiety disorder, including mild to moderate OCD.

   Procedure:
   * Psychologists practicing in the Danish primary sector who have a waiting time of at least four months for psychotherapy treatment will be recruited for the study.
   * The participating psychologists will inform all new clients referred by a GP about the possibility of participating in the trial.
   * Clients who provide written consent will automatically receive the first set of questionnaires.
   * Clients who complete the baseline questionnaires are subsequently randomized to either psychotherapy beginning within two weeks or a waiting list.
   * Clients in either arm of the trial will receive the PHQ-ADS (see Outcome Measures) every other week via an SMS-based solution provided by REDCap.
   * All questionnaires mentioned under the section on "primary and secondary outcome measures" in the section on Outcome Measures are sent out approximately four and a half, eight and a half, and 16 and a half months after the date of the randomization.

   Ethics:
   * The study has been approved by the Institutional Review Board at the Department of Psychology, University of Copenhagen.
   * All data will be stored on drives approved by the Danish Data Protection Authority as appropriately secure, and all rules from the General Data Protection Regulation will be respected.

   Dissemination of Results:
   * The results of the study will be disseminated in at least two scientific articles published in international peer-reviewed journals.
   * In addition, a report will be prepared for the Danish Regions and the Danish Psychological Association, presenting the conclusions of the study and its possible implications for practice.

ELIGIBILITY:
Inclusion Criteria:

Clients:

* All clients who meet the criteria for one of the eleven referral reasons for psychotherapeutic treatment in the Danish primary sector.
* Clients who read and speak proficient Danish to fill in the questionnaires.
* Clients who agree to be randomized through their informed consent.

Psychologists:

* All practicing psychologists employed by the Danish primary sector.
* Psychologists who can commit to the deadlines for beginning treatment.
* Psychologists with at waiting time of approximately four months or longer.

Exclusion Criteria:

- Clients considered unfit for participation or urgently needing psychological or medical help, as determined by the therapist.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 308 (Estimated)
Dates: Start 2025-04-01 (Actual); Primary Completion 2026-10-01 (Estimated); Study Completion 2027-04-30 (Estimated)

PRIMARY OUTCOMES:
Patient Health Questionnaire Anxiety-Depression Scale (PHQ-ADS) | Measured at: Baseline, bi-weekly, four and a half months after randomization date, eight and a half months after randomization date, 12 months after randomization date
  The PHQ-ADS combines the PHQ-9 and the GAD-7 in to a composite measure of depression and anxiety. The PHQ-ADS sums the PHQ-9 and the GAD-7 in to a total score ranging from 0 to 48. The PHQ-ADS has demonstrated high internal reliability as well as convergent validity and con-struct validity in a large sample of primary care patients.

SECONDARY OUTCOMES:
Sheehan Disability Scale (SDS) | Measured at: Baseline, four and a half months after randomization date, eight and a half months after randomization date, 12 months after randomization date
  The SDS is a three-item rating scale that assesses functioning in relation to three domains: work and/or education, social relationships, and family life. The client rates the extent to which a given domain has been impaired by psychological symptoms within the last month, on a scale from 0 ("not at all impaired") to 10 ("very severely impaired").
The WHO-5 well-being index (WHO-5) | Measured at: Baseline, four and a half months after randomization date, eight and a half months after randomization date, 12 months after randomization date
  The WHO-5 is a five-item rating scale on psychological wellbeing. Each item relates to wellbeing within the past two weeks and is rated on a scale from 0 ("none of the time") to 5 ("all of the time"). The total raw score is multiplied by four to compute a percentage scale from 0 (absence of wellbeing) to 100 (maximal wellbeing).
Cohen's Perceived Stress Scale (PSS) | Measured at: Baseline, four and a half months after randomization date, eight and a half months after randomization date, 12 months after randomization date
  The PSS is a ten-item questionnaire assessing the client's experience of stress within the last month. The items are rated on a 5-point Likert scale ranging from 0 ("never") to 4 ("very often"), with a sum score ranging from 0-40.
The Client Satisfaction Questionnaire (CSQ) | Measured at: Baseline, four and a half months after randomization date.
  The CSQ is an eight-item questionnaire assessing the client's satisfaction with the therapy. The items are rated on a four-point Likert scale ranging from one to four, with a sum score ranging from 8-32.
The Negative Effects Questionnaire (NEQ) | Measured at: Baseline and four and a half months after randomization date.
  The NEQ is a 20-item questionnaire assessing the occurrence and severity of a series of negative events associated with receiving psychotherapy.

CONTACTS AND LOCATIONS:
Overall Officials: Stig Poulsen, Professor, Principal Investigator — University of Copenhagen; Ole Karkov Østergård, Associate Professor, Study Chair — Aalborg University; Carsten Hjorthøj, Associate Professor, Study Chair — University of Copenhagen; Celia Faye Jacobsen, PhD, Study Chair — University of Copenhagen
Locations (1):
- University of Copenhagen, Copenhagen, Central Region, Denmark

IPD SHARING:
Plan to Share IPD: No
No participant data is planned to be shared with other researchers besides the EPIC research team members.

REFERENCES:
- See also: The official website for the EPIC trial — https://psy.ku.dk/epic/